CLINICAL TRIAL: NCT02538380
Title: EUS-B-FNA vs EUS-FNA for Left Adrenal Gland Analysis in Lung Cancer
Brief Title: EUS-B-FNA vs EUS-FNA for Left Adrenal Gland Analysis in Lung Cancer Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Prof J.T. Annema, Prof Dr, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NL50139.018.14
Record Dates: First submitted 2015-08-31; First posted 2015-09-02 (Estimated); Last update posted 2015-09-02 (Estimated); Status verified 2015-06

CONDITIONS: Suspected Left Adrenal Gland Metastasis in Lung Cancer
Keywords: Lung cancer; Adrenal gland metastasis
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- EUS-B-FNA for LAG analysis (Experimental): All patients will undergo a mediastinal nodal staging procedure with the EBUS scope (EBUS + EUS-B) (routine clinical care) followed by an evaluation of the LAG including LAG sampling (experimental). Subsequently, all patients undergo a conventional EUS procedure with sampling of the LAG (current standard of care)
  Interventions: Procedure: EUS-B-FNA followed by EUS-FNA for LAG analysis

INTERVENTIONS:
Procedure: EUS-B-FNA followed by EUS-FNA for LAG analysis

SUMMARY:
The purpose of this study is to compare EUS-B-FNA (using the EBUS scope)with EUS-FNA for left adrenal gland analysis in lung cancer patients.

DETAILED DESCRIPTION:
Rationale:

The adrenal glands are a predilection site for distant metastases (M1b) in patients with lung cancer.

However, even in a patient with a confirmed lung cancer an enlarged adrenal lesion is still more likely to be benign than to be malignant(4). Therefore tissue sampling of the left adrenal gland (LAG) is obligatory to either confirm or rule out metastases. Sampling is regularly performed by a transgastric endoscopic approach using a conventional GI-EUS scope. The aim of this study is investigate the success rate of endoscopic ultrasound guided fine-needle aspiration using the EBUS scope (EUS-BFNA) for left adrenal gland analysis in patients with lung cancer and an on imaging suspected left adrenal gland.

Hypothesis:

EUS-B guided transgastric FNA of suspected left adrenal glands (LAG) reduces the need for conventional EUS- FNA by half.

Study design:

A prospective cohort design Setting: international, multicenter

Study population:

Patients with (suspected) lung cancer, an indication for mediastinal nodal staging and a for malignancy suspected LAG on imaging.

Intervention:

All patients will undergo a mediastinal nodal staging procedure with the EBUS scope (EBUS + EUSB) (routine clinical care) followed by an evaluation of the LAG including LAG sampling (experimental). Subsequently, all patients undergo a conventional EUS procedure with sampling of the LAG (current standard of care)

Main study endpoint:

The proportion of patients with a successful EUS-B-FNA procedure for LAG analysis. Successful is defined as: LAG is visible, sampling is possible and adequate material for cytopathological evaluation is obtained. Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Distant metastases of lung cancer like LAG metastases have significant impact on both the prognosis and treatment. In the majority of patients with an indication for LAG sampling by endosonography, there is also an indication for mediastinal nodal tissue sampling. In case both the mediastinal lymph nodes and the LAG can be evaluated with the same scope, patients can be evaluated for nodal and distant metastasis with just a single instead of two separate scopes. This will be beneficial for patients (reduced investigation time) and is additionally cost -effective. So far EUS-B of LAG has been shown to be safe and feasible.

ELIGIBILITY:
Inclusion Criteria:

* (Suspected) Lung Cancer
* For malignancy suspected LAG on imaging (enlarged based on CT and/or FDG avid based on FDG-PET);
* Indication for endosonographic mediastinal staging by EBUS;
* Indication for LAG sampling;

Exclusion Criteria:

* Contraindication for EUS;
* Pregnancy;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2015-03; Primary Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients with a successful EUS-B-FNA procedure for LAG analysis. | within 3 weeks after inclusion
  Successful is defined as: LAG is visible, sampling is possible and adequate material for cytopathological evaluation is obtained.

CONTACTS AND LOCATIONS:
Overall Officials: Jouke T Annema, MD PhD, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (2):
- Netherlands (2):
  - Academic Medical Center, Amsterdam
  - University Hospital Nijmegen, Nijmegen